CLINICAL TRIAL: NCT06373913
Title: The Role of Proprotein-convertase-subtilisin/Kexin-type 9 in Kidney Damage in Nephrotic Syndrom
Acronym: PCSK9
Status: Recruiting | Type: Observational
Sponsor: Kolding Sygehus (Other)
Collaborators: Odense University Hospital (Other); Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MASP2NSRZL
Record Dates: First submitted 2023-10-10; First posted 2024-04-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hyperlipidemias; Nephrotic Syndrome
MeSH Terms: conditions — Hyperlipidemias; Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, blood samples, kidney biopsy tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nephrotic syndrome: Patients with nephrotic syndrome (n=32). Blood samples and 24 hour urine samples will be obtained an all participants. Kidney biopsy will be used from 11 test persons, whos been subjected to kidney biopsy unrelated to the research project.
  3
- Kidney healthy controls: Patient with normal kidney function and no proteinuria (n=32). Blood samples and 24 hour urine samples will be obtained an all participants.
- Kidney biopsy control: Patients without proteinuria who is subjected to kidney biopsy regardless of the research project.

SUMMARY:
Nephrotic syndrome (NS) is characterized by gross proteinuria (>3.5 g/day), hypoalbuminaemia, edema and often hyperlipidemia. Hyperlipidemia is correlated with increased morbidity and mortality.

The study aim is to investigate the role of the protein convertase subtilisin/kexin type 9 (PCSK9) in hyperlipidemia of NS, which has been suggested to play an important role. This is done by testing the following hypotheses:

1. PCSK9 is increased in patients with NS and hyperlipidemia compared to kidney-healthy controls
2. The level of PCSK9 in plasma correlates to the degree of proteinuria.
3. PCSK9 i increased in the kidney tissue of patients with NS

The study will compare plasma levels of PCSK9 in correlation with degree of protein in the urine between test persons with NS and kidney healthy controls. Furthermore the investigators will study the the degree of PCSK9 in the kidney in biopsies obtained from test persons with nephrotic syndrome and test persons without proteinuria.

DETAILED DESCRIPTION:
Hyperlipidemia in kidney disease is associated with a substantially increase of risk in development of atherosclerotic cardiovascular disease (CVD) (European Atherosclerosis Society 2011). Furthermore animal studies have suggested that hyperlipidemia escalates progression of glomerular injury.

Nephrotic syndrome (NS) - the feature of many primary and secondary glomerulopathies - is characterized by gross proteinuria (>3.5 g/day), hypoalbuminaemia, edema and often hyperlipidemia. The protein Convertase subtilisin/kexin 9 (PCSK9) is over expressed in NS and has been suggested to play an important role in developing of hyperlipidemia. PCSK9 increases the LDL receptor degradation by preventing it from recycling to the cell membrane, resulting in increased plasma LDL cholesterol.

PCSK9 is produced primarily in the liver, but to a lesser extent in the brain, intestine and kidney. A recent study found that the expression of renal PCSK9 is increased in mice with experimental NS compared to controls. The investigators want to further explore this.

The overall aim is to decrease morbidity and mortality associated with NS and hyperlipidemia, by testing the following hypotheses:

1. PCSK9 is increased in patients with NS and hyperlipidemia compared to kidney-healthy controls
2. The level of PCSK9 in plasma correlates to the degree of proteinuria.
3. PCSK9 i increased in the kidney tissue of patients with NS

The study want to compare plasma levels of PCSK9 in correlation with degree of protein in the urine between test persons with NS and kidney healthy controls. Furthermore the investigators will study the the degree of PCSK9 in the kidney in biopsies obtained from test persons with nephrotic syndrome and test persons without proteinuria in a subgroup of the test persons assigned to kidney biopsy regardless of the project.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Patients admitted to the Medical Department and/or the Medical Emergency Department, Kolding Sygehus.

Exclusion Criteria:

* Refusal to give informed consent
* Treatment with PCSK9 inhibitors
* Any acute or chronic condition that would limit the ability of the patient to participate in the study
* Control group: proteinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with >3.5 g/day of proteinuria will be included in the nephrotic syndrome group. Control test subjects will be excluded if proteinuria occur.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Plasma PCSK9 correlated to the degree of protein in the urine | Measured at inclusion and for the nephrotic group after remission, if this is accomplished within a year
  PCSK9 in plasma measured by ELISA, correlated to protein in 24hour urine
Degree of PCSK9 in kidney tissue | Measured at inclusion in test person group, if this is performed within in the study period (before august 2028).
  Immunohistochemistry; degree of staining a in test persons, who are subjected to kidney biopsy.

SECONDARY OUTCOMES:
Localization of PCSK9 in kidney tissue | Measured at inclusion in test person group, if this is performed within in the study period (before august 2028).
  Immunohistochemistry; localization of staining a in test persons, who are subjected to kidney biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kolding Sygehus, Lillebælt Hospital, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu S, Vaziri ND. Role of PCSK9 and IDOL in the pathogenesis of acquired LDL receptor deficiency and hypercholesterolemia in nephrotic syndrome. Nephrol Dial Transplant. 2014 Mar;29(3):538-43. doi: 10.1093/ndt/gft439. Epub 2013 Oct 28. PMID 24166456
- [Background] Molina-Jijon E, Gambut S, Mace C, Avila-Casado C, Clement LC. Secretion of the epithelial sodium channel chaperone PCSK9 from the cortical collecting duct links sodium retention with hypercholesterolemia in nephrotic syndrome. Kidney Int. 2020 Dec;98(6):1449-1460. doi: 10.1016/j.kint.2020.06.045. Epub 2020 Aug 1. PMID 32750454
- [Background] Haas ME, Levenson AE, Sun X, Liao WH, Rutkowski JM, de Ferranti SD, Schumacher VA, Scherer PE, Salant DJ, Biddinger SB. The Role of Proprotein Convertase Subtilisin/Kexin Type 9 in Nephrotic Syndrome-Associated Hypercholesterolemia. Circulation. 2016 Jul 5;134(1):61-72. doi: 10.1161/CIRCULATIONAHA.115.020912. PMID 27358438